CLINICAL TRIAL: NCT03083392
Title: Endosseous Oroantral Port for Minimal Intervention in Treating Chronic Sinusitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, ruth angel dar, Principal Investigator, Western Galilee Hospital-Nahariya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0015-17-NHR
Record Dates: First submitted 2017-03-05; First posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Maxillary Sinusitis
Keywords: DIVA; sinusitis; maxillary
MeSH Terms: conditions — Maxillary Sinusitis; Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): treatment of chronic maxillary sinusitis using DIVA system
  Interventions: Procedure: treatment of chronic maxillary sinusitis using DIVA system; Device: "dynamic implant valve approach" - DIVA system

INTERVENTIONS:
Procedure: treatment of chronic maxillary sinusitis using DIVA system — chronic maxillary sinusitis treatment utilizing DIVA system for antral lavage
Device: "dynamic implant valve approach" - DIVA system — The DIVA system will be used to apply saline lavage to the maxillary sinus

SUMMARY:
This study is intended to evaluate the efficiency of utilizing "dynamic implant valve approach" (DIVA) system in treating chronic maxillary sinusitis.

DETAILED DESCRIPTION:
A prospective study aimed to test the efficiency of a minimal interventional approach in treating chronic maxillary sinusitis. The "dynamic implant valve approach" (DIVA), a minimally invasive approach utilizes a dental implant, designed with an internal sealing screw that might serve as drug delivery system via its channel. The implant is inserted to a posterior maxillary edentulous area, creating a connection between the sinus cavity and the oral cavity (Oro-antral connection), hence, provides a controlled working channel for diagnosis and treatment of the disease (e.g; allowing drainage, lavage and sinus endoscopy). The implant is a medical device approved for use at the anatomical area of interest.

The treatment method proposed in this study is based on the principle of a conventional treatment of washing the maxillary sinus cavity called "Antral puncture and lavage".

The changes that are proposed in this study could make the operation more convenient and effective in the therapeutic level, both for the patient and the clinician for the following reasons:

* DIVA (Dynamic Implant Valve Approach) Implant with a multi- useful working channel: the mere presence of the canal in the center of the implant with a screw seal, ensures controlled Oro-antral connection, and enables multiple endoscopy and lavage procedures until resolution of the pathological condition is achieved.
* The anatomical location of the puncture / penetration to the sinus - is performed in the maxillary edentulous region. This is the lowest area of the sinus cavity (standing or sitting posture), which utilizes gravity for drainage and extraction of the contaminated contents of the sinus.

By appropriate advance planning, the implant, after eradication of the disease, can later be used for prosthetic purposes.

ELIGIBILITY:
Inclusion Criteria:

* No medical history of diseases involving bone metabolism
* Unilateral or bilateral maxillary sinusitis, as evident by radiographic and endoscopic modaleties, which have not responded to optimal conservative treatment
* Patient who is edentulous in the maxillary region and is interested in dental implant
* The patient does not participate in another clinical study
* The patient can read and understand the informed consent

Exclusion Criteria:

* Medical history of increased risk of developing bone necrosis (MRONJ - medically related osteonecrosis of the jaw , or ORN - osteoradionecrosis)
* patients who are not interested or need dental implants
* Patients with maxillary sinus neoplastic pathology
* Chronic maxillary sinusitis with polyps
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
resolution of chronic maxillary sinusitis | three months
  After three months of follow-up, the patient will be assessed by a combination of medical tests (clinical, endoscopic and radiologic assessment), in order to determine if the maxillary sinusitis has completely resolved. The investigators expect to see complete resolution of the sinus pathological state (e.g. no evidence of sinusitis)

CONTACTS AND LOCATIONS:
Overall Officials: Samer Srouji, Prof., Study Director — Western Galilee Medical Center
Locations (1):
- Western Galilee Medical Center, Nahariya, Israel

REFERENCES:
- [Background] Albu S, Baciut M, Opincariu I, Rotaru H, Dinu C. The canine fossa puncture technique in chronic odontogenic maxillary sinusitis. Am J Rhinol Allergy. 2011 Sep-Oct;25(5):358-62. doi: 10.2500/ajra.2011.25.3673. PMID 22186252
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Background] Ludlow JB, Ivanovic M. Comparative dosimetry of dental CBCT devices and 64-slice CT for oral and maxillofacial radiology. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Jul;106(1):106-14. doi: 10.1016/j.tripleo.2008.03.018. Epub 2008 May 27. PMID 18504152
- [Background] Nahlieli O, Moshonov J, Zagury A, Michaeli E, Casap N. Endoscopic approach to dental implantology. J Oral Maxillofac Surg. 2011 Jan;69(1):186-91. doi: 10.1016/j.joms.2010.07.071. Epub 2010 Nov 2. PMID 21050639
- [Background] Nahlieli O, Casap N, Moshonov J, Zagury A, Michali E, Samuni Y. A novel dental implant system with an internal port for endoscopic closed sinus augmentation: a feasibility study in pigs. Int J Oral Maxillofac Implants. 2013 Nov-Dec;28(6):e556-61. doi: 10.11607/jomi.te36. PMID 24278950
- [Background] Neugebauer J, Ritter L, Mischkowski RA, Dreiseidler T, Scherer P, Ketterle M, Rothamel D, Zoller JE. Evaluation of maxillary sinus anatomy by cone-beam CT prior to sinus floor elevation. Int J Oral Maxillofac Implants. 2010 Mar-Apr;25(2):258-65. PMID 20369083
- [Background] Rosenfeld RM, Andes D, Bhattacharyya N, Cheung D, Eisenberg S, Ganiats TG, Gelzer A, Hamilos D, Haydon RC 3rd, Hudgins PA, Jones S, Krouse HJ, Lee LH, Mahoney MC, Marple BF, Mitchell CJ, Nathan R, Shiffman RN, Smith TL, Witsell DL. Clinical practice guideline: adult sinusitis. Otolaryngol Head Neck Surg. 2007 Sep;137(3 Suppl):S1-31. doi: 10.1016/j.otohns.2007.06.726. PMID 17761281